CLINICAL TRIAL: NCT01892072
Title: VEGF Signaling Promotes Cell Growth and Metastasis in Hepatocellular Carcinoma in a VEGF Receptor Mediated Pathway
Acronym: HCC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Guangdong Province, Department of Science and Technology (Other Government)
Responsible Party: Principal Investigator, Ming Kuang,MD,PhD, MD,PhD, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: k0113011-2013VEGF
Record Dates: First submitted 2013-06-30; First posted 2013-07-03 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; HCC; VEGF signaling pathway
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cut tissue into small pieces (~2 mm2)and wash in drops of saline (1x PBS). Place pieces individually into LN2 in Styrofoam cup. Transfer pieces into LN2-cooled 1.5 mL cryovial. Pour out excess LN2 from vial, then seal and keep in LN2 until freezer storage.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCC patients: Hepatocellular carcinoma patients treated by surgical treatment
  Interventions: Procedure: surgical treatment

INTERVENTIONS:
Procedure: surgical treatment — all the patients in the study must have been treated by the surgery at the first time and have been confirmed as 'complete section' by the post-surgery radiological image.

SUMMARY:
The investigators study the VEGF signaling in HCC cell lines and its mechanism in HCC growth, proliferation and apoptosis.

DETAILED DESCRIPTION:
Several studies have documented the elevated expression of VEGF, VEGFR1 and VEGFR2 in HCC cell lines and tumor tissues. Another study observed a sequential elevation of VEGF in low-grade dysplasia, high-grade dysplasia and early stage HCC. Clinical analyses have discovered the high expression of VEGF is correlated with tumor progression, vascular invasion, distal metastasis and poor prognosis. However, few studies have been conducted to investigate the VEGF signaling in HCC cells and its possible mechanism in regulating HCC growth.Therefore,we try to clarify the mechanism of VEGF signal in HCC growth,proliferation and apoptosis.

ELIGIBILITY:
Inclusion Criteria:

1. hepatocellular patients diagnosed through biopsy;or either dynamic imagine with a diagnosis of hepatocellular carcinoma and alphafetoprotein>400μg/L；or two or more dynamic imagine with a diagnosis of hepatocellular carcinoma
2. Child-Pugh A or B
3. well preserved renal and hematopoietic Function
4. receive surgical therapy
5. achieve complete section accessed by contrast-enhanced CT

Exclusion Criteria:

1. incomplete section
2. remote metastasis
3. Child-Pugh C
4. combination with other hepatobiliary disease
5. suffer from other tumors concurrently or in last five years

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hepatocellular carcinoma patients underwent surgical therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
the variation of the quantity of VEGF signal pathway genes in normal liver tissue,peri tumor,tumor and metastasis. | the day when conducting surgery (day 1)
  the sections would be collected as previously described.Western blot,immunohistochemistry,PCR would be conducted to find out the variation between the normal liver tissue and tumor,tumor and meta(if have).

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, MD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China